CLINICAL TRIAL: NCT07329114
Title: Prospective, Unblinded, Randomized, Controlled Investigation to Evaluate the Clinical Efficacy of PowerHeal™ Bioelectric Bandage in Managing Infected Traumatic Wounds
Brief Title: Healing Electroceutical Dressing for the Recovery of Open Wounds (HERO)
Acronym: HERO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chandan Sen (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor-Investigator, Chandan Sen, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY25010029; MTEC-24-01-MPA-085 (Other: The Medical Technology Enterprise Consortium, Inc. (MTEC))
Record Dates: First submitted 2026-01-07; First posted 2026-01-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Wound Heal; Wound Infection; Wound Healing Delayed; Wound of Skin; Infections
Keywords: bandage
MeSH Terms: conditions — Wound Infection; Infections

STUDY DESIGN:
Intervention Model Description: How well the PowerHeal™ Bioelectric Bandage-a special wireless bandage that uses gentle electrical signals-helps heal infected wounds caused by injuries, will be tested. The study will take place at a minimum of three medical sites in Ukraine, with support and training from experts in the United States at the University of Colorado and the University of Pittsburgh. All teams will stay in close contact throughout the study. This international collaboration aims to find out if this new type of bandage can reduce infections and speed up healing for people with serious wounds.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care (SOC) Group (Active Comparator): The choice of wound dressing and timing of dressing changes will be determined by the investigation doctor until the participant's wound heals, or until the participant is discharged.
  Interventions: Device: Standard of care dressing
- SOC + PowerHeal™ Bioelectric Bandage Group (Experimental): * The first SOC + PowerHeal™ Bioelectric Bandage will be applied within 24 hours of randomization.
  * Each participant is expected to need at least 15 PowerHeal™ Bioelectric Bandages throughout the study.
  PowerHeal™ Bandage Change Schedule
  Dressing change frequency depends on how much fluid (exudate) the wound produces.
  * Day 0-7 and Day 7-14: Minimum of 2 times per week, up to every other day.
  * Day 14-28: Minimum of once per week, more as needed dependent on wound exudate.
  Interventions: Device: PowerHeal™ Bioelectric Bandage; Device: Standard of care dressing

INTERVENTIONS:
Device: PowerHeal™ Bioelectric Bandage — PowerHeal™ Bioelectric Bandage is a flexible fabric electroceutical based wound bandage offering ease of portability with long shelf life and stable for storage under any conditions. PowerHeal™ Bioelectric Bandage may be preventively used on fresh wounds. PowerHeal™ Bioelectric Bandage can directly disrupt the biofilm infection and enhance host resilience such as restoring skin barrier function (10). Productive management of bacterial biofilm/MDR infection or risk of such infection will minimize healing complications. This will result in fewer treatments and corrective procedures and earlier return to daily life for patients with traumatic wounds/burns.
  Other Names: wireless electroceutical dressing (WED)
  Arms: SOC + PowerHeal™ Bioelectric Bandage Group
Device: Standard of care dressing — SOC will be determined by local established guidelines and participant needs. This may include sutures, staples, liquid skin adhesives, adhesive surgical tape, gauze dressings and negative pressure wound therapy treatment strategies.

SUMMARY:
The goal of this clinical trial is to determine whether the wireless electroceutical dressing (WED) called PowerHeal™ Bioelectric Bandage, improves care of infected wounds by clearing the infection and helping the wound heal better.

The main hypotheses it aims to answer are:

1. WED promotes wound closure, as determined by wound area measurement
2. WED manages wound infection in civilian and military wounds in Ukraine, as determined by clinical assessment of wound infection by measuring the numbers and types of relevant microbes.

Researchers will compare to see if PowerHeal™ Bioelectric Bandage the dressing used in the SOC group

Participants will get their dressings changed per the protocol, wound image and swab will be taken.

DETAILED DESCRIPTION:
Managing bacterial burden is necessary for effective wound healing. Military wounds are severely complex due to rise in multidrug resistant bacterial infections. A FDA cleared commercially available disposable, wireless electroceutical dressing fabric is able to generate a low electric field in presence of exudate in the wound environment. The electric field, along with the micro-molar amounts of superoxide anion radicals that is generated in the wound microenvironment, initiate a bactericidal and a pro-healing signaling cascade resulting in improved wound healing without the encumbrance of a bulky dressing.

There will be five visits over the course of 28 ± 2 days. Participants will be randomized and divided into two groups: one group will receive the standard of care (SOC) dressing and the other will receive the bioelectric bandage. Dressing change intervals will depend on the group the participant randomized to and how exudating the wound is.

The investigation doctor will collect demographic data - such as, age, sex, race; general medical history, and targeted wound data -such as cause, size, location, duration and total number of traumatic wounds. Standard of care clinical lab results (complete blood count, liver and kidney functions, presence and level of inflammation) will also be collected to evaluate body functions and health status . No blood will be collected for this study.

Vital signs (body temperature, respiratory rate, heart rate, blood pressure, level of oxygen in blood) will be measured. The doctor will also look for signs of wound infection (of the investigation wound) including, redness, warmth, swelling, drainage, discoloration, friable granulation, foul odor, necrosis, and pustule/vesicles/boils. Participants will be asked about their pain experience compared to the moment of the injury.

A swab of the investigation wound will be collected per standard study guidelines at each investigation timepoint (unless the wound heals). A member of the study team will clean the wound using sterile sodium chloride solution, then gently rotate a sterile swab over a small area of the wound to collect a sample. All collected wound swabs will be sent to and processed in a central lab within Ukraine to check the infection status of the wound. Microbes detected in the wound will then be further analyzed in a separate central laboratory in the US to look at important factors such as antibiotic resistance. The results of the research wound swabs and analysis data will not be shared with the participant, or their medical care provider.

At each investigation timepoint, the investigation wound will also be photographed by the investigator or a member of the investigation team using the camera function on a standard smartphone to see if there is any change before and after receiving the treatment. The investigation wound will also be measured for size by holding a clear, sterile, wound measurement tool on top of the wound.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male participants 18-105 years of age
2. Hospital admission (or boarding in an emergency department or other area awaiting hospital admission) at participating clinical sites in Ukraine
3. At least one infected traumatic wound(s) between 20-40 cm2 in size. Probable or confirmed wound infection(s) will be determined by on-site physicians' clinical judgment and the presence of two or more of the following clinical indicators of wound infection:

   1. Presence of worsening pain (from the moment of injury)
   2. Erythema (redness)
   3. Warmth (heat)
   4. Edema (swelling)
   5. Purulent exudate (drainage)
   6. Delayed healing
   7. Discoloration
   8. Friable granulation
   9. Foul odor
   10. Wound margin breakdown or necrosis with or without fever
   11. Pustules, vesicles, boils
4. Participant or legal representative provides written informed consent prior to investigation procedures
5. Participant understands and agrees to adhere to planned investigation procedures

Exclusion Criteria:

1. Allergy to silver or zinc
2. Women who are pregnant or nursing
3. Women of childbearing potential without a documented negative pregnancy test during the current hospitalization or women of childbearing potential who refused pregnancy testing during screening
4. Sponsor or contract research organization (CRO) staff directly involved in the conduct of the investigation, and site staff supervised by the investigator, and their respective family members
5. > 60 days from the initial traumatic injury
6. Known prisoner
7. The patient is expected to be discharged from the hospital within the next 24 hours
8. Medical condition other than the acute traumatic wound (and its manifestations) that is likely to result in death within 14 days of randomization
9. Moribund condition, defined as life expectancy less than 48 hours from randomization
10. Patients undergoing comfort care measures only such that treatment focuses on end-of-life symptom management over prolongation of life
11. Expected inability or unwillingness to participate in study procedures
12. In the opinion of the investigator, participation in the investigation is not in the best interest of the patient

Note: Allergies to parabens and acrylates will also be considered. While they are not direct exclusions, participants with these allergies should avoid being enrolled.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
change in wound area | 28 days (± 2 days)
  Assess the efficacy of WED in promoting wound closure.
  The digital photos taken at all visits will be quantitatively evaluated using ImageJ software that can measure the wound area. These measurements will be used for detailed analysis of wound closure over the period of study. Percentage decrease in wound area compared to SOC - from baseline (day 0) to final visit (day 28,± 2 days) will be calculated and analyzed, thus comparing range and rate of change between the two groups SOC and SOC + PowerHeal™ Bioelectric Bandage in aggregate.
  Adjustment for the correlated variance due to repeated measures will be made throughout the analysis. All analysis will be conducted at 0.05 level of significance.

SECONDARY OUTCOMES:
Change in microbial population - types of strains and numbers of colonies | 28 days (± 2 days)
  Assess the efficacy of PowerHeal™ Bioelectric Bandage in wound infection management.
  Swabs will be collected per standard local study guidelines. Clearance or presence of the numbers and types of clinically relevant microbes such as multidrug resistant (MDR) strains of ESKAPE pathogens (Enterococcus faecium, Staphylococcus aureus, Klebsiella pneumoniae, Acinetobacter baumannii, Pseudomonas aeruginosa, Enterobacter spp.), Candida auris, and all Gram-negative isolates of clinical concern (e.g. Serratia sp., Citrobacter sp.) will be determined to evaluate the change in microbial load. Clinical assessments of wound infection will be calculated and compared across baseline, Day 7 (± 2 days), Day 14 (± 2 days) and end of study samples.
  The speciation provided by the laboratory conducting the analysis will determine changes in microbial pathogen over time. Adjustments will be made for variances due to repeated measures, and all analyses will be conducted at 0.05 level of significance.

CONTACTS AND LOCATIONS:
Overall Officials: Chandan K. Sen, PhD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- Ivano-Frankivsk Central Clinical Hospital, Ivano-Frankivsk, Ivano-Frankivsk Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schultze T, Hogardt M, Velazquez ES, Hack D, Besier S, Wichelhaus TA, Rochwalsky U, Kempf VA, Reinheimer C. Molecular surveillance of multidrug-resistant Gram-negative bacteria in Ukrainian patients, Germany, March to June 2022. Euro Surveill. 2023 Jan;28(1):2200850. doi: 10.2807/1560-7917.ES.2023.28.1.2200850. PMID 36695452
- [Background] Banerjee J, Das Ghatak P, Roy S, Khanna S, Sequin EK, Bellman K, Dickinson BC, Suri P, Subramaniam VV, Chang CJ, Sen CK. Improvement of human keratinocyte migration by a redox active bioelectric dressing. PLoS One. 2014 Mar 3;9(3):e89239. doi: 10.1371/journal.pone.0089239. eCollection 2014. PMID 24595050
- [Background] Banerjee J, Das Ghatak P, Roy S, Khanna S, Hemann C, Deng B, Das A, Zweier JL, Wozniak D, Sen CK. Silver-zinc redox-coupled electroceutical wound dressing disrupts bacterial biofilm. PLoS One. 2015 Mar 24;10(3):e0119531. doi: 10.1371/journal.pone.0119531. eCollection 2015. PMID 25803639